CLINICAL TRIAL: NCT03520062
Title: The Effect of Liraglutide on Pancreatic Hormones and Its Size
Acronym: LIRAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolai Jacob Wewer Albrechtsen (Other)
Collaborators: Hvidovre University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Nicolai Jacob Wewer Albrechtsen, Postdoc, MD, PhD, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LIRAP
Record Dates: First submitted 2018-04-24; First posted 2018-05-09 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Obesity
Keywords: Amylase; Lipase; GLP-1
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GLP-1 Receptor Agonist (Liraglutide) (Experimental): 3.0mg daily dose
  Interventions: Drug: Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml

INTERVENTIONS:
Drug: Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml — Treatment with Liraglutide (3.0mg per day) for ~6 weeks

SUMMARY:
Glucagon-like peptide-1 (GLP-1) is a gastrointestinal hormone used to treat type 2 diabetes and severe overweight (Liraglutide).The two pancreas enzymes: amylase and lipase are slightly elevated in GLP-1 treated compared with placebo-treated individuals. Increased levels of these two enzymes (amylase and lipase) are associated with acute inflammation of the pancreas (acute pancreatitis). In humans treated with GLP-1 (receptor agonist) there have not been found an increased risk of acute pancreatitis.

Animal and cell studies have shown that the increased levels of amylase and lipase in the blood are not due to an inflammatory state but adaptive changes (volume increase) of the pancreas.

The investigators (professor Jens Juul Holst, professor Sten Madsbad) want to investigate whether the increased levels of amylase and lipase in the blood of individuals treated with the GLP-1 analogue Saxenda are due adaptive changes of the pancreas. This will be achieved by measuring amylase and lipase before, during and after treatment with a GLP-1 receptor agonist, and at the same time use advanced scanning equipment (PET-MR) from the Clinical Physiological and Nuclear Medical Department at Rigshospitalet, which can determine any volumetric changes in the pancreas with high reproducibility.

The scan will be centered on the pancreas, other organs are not evaluated why the study is not designed to detect any malignant findings in the pancreas or other organs.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 26 og < 50 kg/m2

Exclusion Criteria:

* Abdominal Diameter >60cm type 1 or type 2 diabetes Heart Failure or Disease Statins Kidney or Liver disease Thyroid Disease Inflammatory Bowel Disease Gastroparesis Cancer Lung disease Psychiatric disease Gastric Bypass operation Previous pancreatitis Increased alcoholic consumption Familiar incidence of multiple endocrine neoplasia Previous treatment with GLP-1 (incretin) based medicine Pacemaker or other non-MR-compatible devices

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Volumetric Changes of the Pancreas | 6 weeks
  Measurements of the pancreas volumen using magnetic resonance imaging-positron emission tomography based technology

SECONDARY OUTCOMES:
Changes in Plasma Concentrations of Pancreatic Amylase and Lipase | 6 weeks
Changes in body weight | 6 weeks
Changes in glycemic index | 6 weeks
Plasma concentrations of glucagon, insulin and citrullin | 6 weeks
Plasma concentrations of the drug | 6 weeks
Other MR based changes in the pancreas (edema, cellularity and structural changes) | 6 weeks
Uptake of fluorothymidine tracer in the pancreas measured by PET | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
We have yet not decided to share IPD as this also would require approval from the ethical and data approval comite